CLINICAL TRIAL: NCT03372811
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Controlled, Two-Center, Phase 2b Clinical Trial to Evaluate the Efficacy and Safety of TC Cream In Treating Patients With Psoriasis Vulgaris.
Brief Title: Efficacy and Safety of TC Cream In Treating Patients With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Psoriasis Research Institute of Guangzhou (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105883-1
Record Dates: First submitted 2017-11-30; First posted 2017-12-14 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TC cream (10%) (Active Comparator)
  Interventions: Drug: TC cream
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: TC cream — A well-characterized botanical drug for topical treatment of psoriasis vulgaris
  Arms: TC cream (10%)
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Parallel-Controlled, Two-Center, Phase IIb Clinical Trial to Evaluate the Efficacy and Safety of TC cream In Treating Patients with Psoriasis Vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-70 years old. Both men and women and members of all races and ethnic groups
* Consistent with diagnostic criteria of stable phase psoriasis vulgaris and have at least two target lesions suitable for evaluation
* Women of childbearing age must be using birth control strategies defined by one of the following: 1) a barrier method (condom) and/or 2) oral contraceptives, during the 8-week study period.
* ISGA score ≥ 2 (at least mild severity)
* BSA (stable stage group): 1%≤ to ≤20%
* Signed a written informed consent document
* No additional exposure to the sun

Exclusion Criteria:

* Subjects in pregnancy, preparing for pregnancy or breast feeding
* History of hyperergic or photosensitivity
* History of complicated cardiovascular diseases, cerebrovascular diseases, severe primary diseases of hepatic, kidney and hematopoietic system, or patients with psychiatric disorders
* History of photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosa
* Within 4 weeks prior to randomizations, patients have taken treatment with following approved or investigational psoriasis therapies on the target lesions:

  * Topical treatments
  * PUVA, UVB or Grenz ray therapy.
  * Any systemic treatments other than biologicals with a possible effect on psoriasis (e.g., corticosteroids, vitamin D analogues, hydroxycarbamide, azathioprine, methotrexate, cyclosporine, other immunosuppressant).
  * Any types of other investigational therapies for psoriasis
* Within 3 months prior to randomizations, patients have taken systemic treatments with retinoids or biological therapies (marketed or otherwise) with a possible effect on psoriasis (e.g., alefacept, efalizumab, etanercept, infliximab).
* Planned initiation of, or changes to, concomitant medications that could affect psoriasis (e.g., beta blockers, anti-malaria drugs, lithium) during the double-blind phase of the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic compositions to Coumarins.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Investigator's Static Global Assessment Scale (ISGA) scores of target lesions | up to 12 weeks
  ISGA is a static measurement of the psoriasis status performed by physicians. A 6-point ordinal scale from 0 (minimum) to 5 (maximum) is used for estimation with 0 representing completely clear and 5 for very severe. An ISGA score improvement of ≥2 from baseline is considered an improved outcome.

SECONDARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) scores | up to 12 weeks
  PASI is the most extensively used tool to measure severity of psoriasis by combing the severity of lesions (erythema, induration and desquamation) and affected area into one single score. Scale ranges from 0 (no disease) to 72 (maximal disease)
Change in Dermatology Life Quality Index (DLQI) scores | up to 12 weeks
  DLQI is calculated by summing the score of all questions in questionnaire to measure the impact of psoriasis on the quality of life of a patient. The score ranges from 0 (minimum) to 30 (maximum) with lower scores associated with a better quality of life.
Change in Psoriasis Disability Index questionnaire (PDI) scores | up to 12 weeks
  PDI is used to quantify the impact of psoriasis on quality of patients' daily life. The scale ranges from 0 (minimum) to 90 (maximum) with higher scores indicating impaired quality of life.

OTHER OUTCOMES:
Drug-related incidence and severity of adverse events | week 8
  Percentage of patients with incidence and adverse events related to treatment
Percentage of patients with drug-related changes in clinical laboratory results from baseline | week 8
  Urinalysis laboratory assessments
Percentage of patients with abnormal changes in clinical laboratory results from baseline | week 8
  Biochemistry laboratory assessments
Percentage of patients with drug-related changes in clinical laboratory results from baseline | week 8
  Hematology and coagulation laboratory assessments
Percentage of patients with drug-related changes in physical examination from baseline related to treatment | week 8 and week 12
  Systolic/diastolic blood pressure assessments
Percentage of patients with drug-related changes in physical examination from baseline related to treatment | week 8 and week 12
  Pulse rate assessments
Percentage of patients with drug-related changes in physical examination from baseline related to treatment | week 8 and week 12
  Respiration rate assessments
Percentage of patients with drug-related changes in physical examination from baseline related to treatment | week 8 and week 12
  Body temperature assessments
Percentage of patients with drug-related changes in liver functions from baseline | week 8
  Laboratory assessments of liver functions
Percentage of patients with drug-related changes in renal functions from baseline | week 8
  Laboratory assessments of renal functions
Percentage of patients with drug-related changes in electrocardiography (ECG) from baseline | week 8
  Assessments of PR/PQ intervals, QRS duration and QT intervals

CONTACTS AND LOCATIONS:
Overall Officials: Edward Heilman, MD, Principal Investigator — Department of Dermatology, State University of New York; Peter J. Jenkin, MD, Principal Investigator — Dermatology Associates; Jiang Yang, Ph.D., Study Director — Psoriasis Research Institute of Guangzhou; Liping Yang, MD, Study Chair — Psoriasis Research Institute of Guangzhou
Locations (2):
- United States (2):
  - Department of Dermatology, State University of New York, Downstate Medical Center, New York, New York
  - Dermatology Associates, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No